CLINICAL TRIAL: NCT05271188
Title: Infiltration of Local Anesthetic in the Interspace Between the Popliteal Artery and Capsule of the Posterior Knee "IPACK Block" Versus Adductor Canal Block "ACB" for Pain Relief After Open Wedge High Tibial Osteotomy
Brief Title: IPACK Block Versus Adductor Canal Block in High Tibeal Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salwa Hussein Ahmed Hussein, Assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pain control
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two groups of people who are undergoing open wedge high tibeal osteotomy aged between 40 and 60 yrs old not diabetic and neurologically free
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 who will receive IPACK block (Active Comparator): This group of patients will receive IPACK block immediately before spinal anaesthesia then follow up for 24 hrs to register first pain sensation and analgesic requirements
  Interventions: Procedure: Infiltration of local anaesthetic between popliteal artery and posterior knee capsule
- Group 2 who will receive adductor canal block (Active Comparator): This group of patients will receive adductor canal block immediately before spinal anaesthesia then follow up for 24 hrs to register first pain sensation and analgesic requirements
  Interventions: Procedure: Infiltration of local anaesthetic between popliteal artery and posterior knee capsule

INTERVENTIONS:
Procedure: Infiltration of local anaesthetic between popliteal artery and posterior knee capsule — Adductor canal block (ACB) is a popular peripheral nerve block that has been shown to decrease pain significantly and thereby opioid consumption with minimal effect on quadriceps function [8]. Though ACB provides analgesia to the peripatellar and intra-articular aspect of knee joint, it does not relieve posterior knee pain which is moderate to severe in intensity [9, 10]. The recent technique of an ultrasound (US)-guided local anesthetic infiltration of the interspace between popliteal artery and the capsule of posterior knee (IPACK) has shown to provide significant posterior knee analgesia without affecting the common peroneal nerve (CPN) [11]. We postulated that IPACK will provide better pain relief and improve knee function in the immediate postoperative period compared to ACB
  Other Names: Adductor canal block

SUMMARY:
A comparison between IPACK block and adductor canal block in post operative pain management

DETAILED DESCRIPTION:
Two groups of patients between 40 and 60 yrs who are undergoing open wedge high tibeal osteotomy Group 1 will receive IPACK block with 15 ml Bupivacaine, immediately before spinal anaesthesia .

Group 2 will receive adductor canal block ,also with 15 ml Bupivacaine. before spinal anaesthesia. register the time of first pain sensation and firs IV analgesic dose required in each group

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 - 60 years.
2. American Society of Anesthiologist class ( ASA) I - III
3. BMI 18-35 kg/m2
4. Scheduled for primary unilateral open wedge high tibial osteotomy

Exclusion Criteria:

1. Known allergy to local anesthetics
2. Contraindication to local anesthetics injection e.g. infection at the site of injection
3. Contraindication to spinal anesthesia e.g. coagulopathy.
4. Patients with pre-existing motor or sensory deficits in lower extremities.
5. Insulin or noninsulin dependent diabetes mellitus.
6. systemic corticosteroid use within 30-days of surgery
7. difficulties in comprehending visual analog scale (VAS) pain scores
8. history of arrhythmia or seizures
9. severe renal insufficiency

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
the time of first pain sensation requiring analgesia | 24 hours
  If intervention which is adductor canal block or lPACK block is effective in postoperative pain control that can decrease the lV analgesic agents

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Hussein, Lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No